CLINICAL TRIAL: NCT07064031
Title: Effects of Post Isometric Relaxation and Janda's Approach on Pain, Muscle Endurance and Disability in Patient With Shoudler Girdle Crossed Syndrome
Brief Title: Effects of Post Isometric Relaxation and Janda's Approach in Patient With Shoudler Girdle Crossed Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/24/0144 Muqaddas
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Upper Crossed Syndrome
Keywords: Muscle strength; Muscle Endurance; pain; posture
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus; Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post isometric relaxation (Experimental): This Group Will Receive Post isometric relaxation and Janda . PIR will be perform on upper trapezius and pectorals major muscle. In Janda technique weak muscles will be Strengthened and Tight muscles will be stretched.
  Interventions: Other: Neck Isometrics , TENS and Hot pack
- Janda Technique (Active Comparator): This group is control group and receive only Janda Technique as mentioned weak muscles i.e. serratus Anterior and Rhomboids are strengthened by isometric contraction of these muscles. Stretching of tight muscles i.e. upper trapezius and Pectoralis major muscle.
  Interventions: Other: Neck Isometrics , TENS and Hot pack

INTERVENTIONS:
Other: Neck Isometrics , TENS and Hot pack — Hot apck and TENS applied for 10min each. Using the same amount of light pressure, gently push your head into your hand as you did before. This time, allow the head to move slowly toward the shoulder against the pressure of the hand. This too can be repeated on the opposite side, forwards, backward, and into left and right rotation

SUMMARY:
Shoulder girdle crossed syndrome referred as upper crossed syndrome. In this syndrome, tightness of the upper trapezius and levator scapula on the dorsal side crosses with tightness of the pectoralis major and minor. Weakness of the deep cervical flexors, ventrally, crosses with weakness of the middle, lower trapezius and Rhomboids. Janda Approach treatment involves steps i.e Normalize the Periphery, Restore Muscle Balance, Increase afferent input to facilitate reflexive stabilization and increase endurance in muscles.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial and will be conducted in Riphah Rehabilitation Clinic Lahore. Non-probability convenient sampling will be used to collect the data. Sample size of 54 subjects with age group between 18-50 years will be taken. Data will be collected from the patients having present complaint of neck pain. Outcome measures will be taken using Numeric pain rating scale (NPRS) for pain, Neck disability index (NDI) for disability and Muscle Endurance tests for neck flexors, extensors and lateral flexors, an informed consent will be taken. Subjects will be selected on the basis of inclusion and exclusion criteria and will be equally divided into two groups by random number generator table. Both the Groups will receive Janda treatment as standard physical therapy, while Group A will receive janda's Technique and Muscle Energy Technique. In Janda technique weak muscles will be Strengthened and Tight muscles will be stretched. While group B is control group and receive only Janda Technique. Outcome measures will be measured at baseline and after 4 weeks. Data analysis will be done by SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 18 and 50 years (defined as pain in the area of the neck could be provoked by mechanical characteristics, including sustained neck postures, cervical movement, or manual palpation of the cervical musculature)

Exclusion Criteria:

* Cervical radiculopathy
* History of whiplash injury
* History of cervical and thoracic spine surgery
* Neck pain associated with vertigo

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | upto 4 weeks
  The Numeric Pain Rating Scale (NPRS) is perhaps the most frequently applied scale used to quantify pain intensity in the clinical setting. It is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable
Neck Disability Index (NDI) | upto 4 weeks
  The Neck Disability Index (NDI) is a validated 10-item-questionnaire for the assessment of neck pain. The items of the questionnaire assess deficits in physical and social functioning as well as pain and everyday activities.
Endurance Tests | upto 4 weeks
  Endurance Tests:
  Research by Parazza et al 2014 found the following results when looking at neck endurance strength in flexion and extension:
  Neck flexion: 44 seconds and Neck extension: 261 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Ittefaq Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mubeen I, Malik S, Akhtar W, Iqbal M, Asif M, Arshad A, et al. Prevalence of upper cross syndrome among the medical students of University of Lahore. International journal of Physiotherapy. 2016;3(3):381-4.
- [Background] Dhage P, Anap D. Prevalence of an "Upper Crossed Syndrome in Physiotherapy College Students"-A Cross-Sectional Study. VIMS Health Science Journal. 2019;6(1):10-3.
- [Background] Kage V, Putti B. Effectiveness of stretching and strengthening exercises (Janda's approach) in subjects with postural backache: A randomized controlled trial. Int J Physiother Res. 2015;3(6):1301-6.
- [Background] Bae WS, Lee HO, Shin JW, Lee KC. The effect of middle and lower trapezius strength exercises and levator scapulae and upper trapezius stretching exercises in upper crossed syndrome. J Phys Ther Sci. 2016 May;28(5):1636-9. doi: 10.1589/jpts.28.1636. Epub 2016 May 31. PMID 27313388
- [Background] Guanche C, Knatt T, Solomonow M, Lu Y, Baratta R. The synergistic action of the capsule and the shoulder muscles. Am J Sports Med. 1995 May-Jun;23(3):301-6. doi: 10.1177/036354659502300308. PMID 7661256
- [Background] Umphred D, Byl N, Lazaro R, Roller M. Interventions for neurological disabilities. Neurological rehabilitation. 2001;4:56-134.
- [Background] Sherrington C. On reciprocal innervation of antagonistic muscles. Proc R Soc London B. 1905;76:161-269.
- [Background] El Laithy MH, Fouda KZ. Effect of post isometric relaxation technique in the treatment of mechanical neck pain. Physical Therapy and Rehabilitation. 2018;5(1):20.